CLINICAL TRIAL: NCT05465967
Title: A Comparative Study Between Two Approaches of Ultrasound-Guided Transmuscular Quadratus Lumborum Block on Post-Operative Analgesia After Total Hip Arthroplasty
Brief Title: Transmuscular Quadratus Lumborum Block on Post-Operative Analgesia After Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Abdelhaleem Kamal Nida, assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL block on hip arthroplasty
Record Dates: First submitted 2022-07-07; First posted 2022-07-20 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Quadratus Lumborum Block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: Control Group (Sham Comparator): Patients in this group will receive ipsilateral sham ultrasound-guided block via subcutaneous injection of 1 ml of normal saline after surgery.
  Interventions: Procedure: Quadratus lumborum Block
- Group II:( transverse trans muscular Quadratus lumborum group). (Active Comparator): patients in this group will receive an ipsilateral single-shot of paraspinous sagittal approach of Quadratus lumborum BLOCK(30 ml of plain bupivacaine 0.25%) after surgery using ultrasonographic guidance.
  Interventions: Procedure: Quadratus lumborum Block
- Group III : paraspinous sagittal approach of Quadratus lumborum BLOCK (Active Comparator): patients in this group will receive an ipsilateral single-shot of paraspinous sagittal approach of Quadratus lumborum BLOCK (30 ml of plain bupivacaine 0.25%) after surgery using ultrasonographic guidance.
  Interventions: Procedure: Quadratus lumborum Block

INTERVENTIONS:
Procedure: Quadratus lumborum Block — 1-Transverse transmuscular Quadratus lumborum block: ultrasound transducer will placed transverse to the abdominal flank to visualise abdominal muscle layers. moving the probe posteriorly, the transverse process of the lumbar vertebra, Quadratus lumborum, Psoas Major and erector spinae muscles identified as a 'Shamrock sign'. the needle will inserted through the back muscles to fascial plane between the Quadratus lumborum and Psoas Major, local anesthetic will injected .2- paraspinous sagittal Quadratus lumborum block: ultrasound transducer will be directed caudally in a sagittal plane lateral to the spinous process of L4. moving laterally until the Quadratus lumborum is evident in its long axis with a characteristic sonographic image of three muscle layers appearing from posterior to anterior as: erector spinae, Quadratus lumborum, and Psoas major muscle the needle will be advanced through the muscles, until it pierces the Quadratus lumborum. local anesthetic will be injected.

SUMMARY:
The aim of this study is to compare between the post-operative analgesic effect of two approaches of transmuscular quadratus lumborum block (transverse versus paraspinous sagittal transmuscular QLB) in total hip replacement surgery.

DETAILED DESCRIPTION:
During the preanesthetic assessment, all patients will be educated about the visual analogue scale (VAS) for pain assessment, with scores ranging from 0 to 10 (0 represent no pain, while10 represent maximum intolerable pain).

The patients will be randomly classified into three equal groups (25 patients each). Group allocation will be done by computer generated random numbers and closed opaque sealed envelopes. The study will be designed to be double blind as all patients and postoperative assessor will be blinded to group assignment.

Patients will be randomized to one of three equal groups:

* Group I: Control group (n= 25 patients): Patients in this group will receive ipsilateral sham ultrasound-guided block via subcutaneous injection of 1 ml of normal saline after surgery.
* Group II (n= 25 patients): Patients in this group will receive an ipsilateral single shot of transverse transmuscular approach of QLB (30 ml of plain bupivacaine 0.25%) after surgery using ultrasonographic guidance.
* Group III (n= 25 patients): patients in this group will receive an ipsilateral single-shot of paraspinous sagittal approach of QLB (30 ml of plain bupivacaine 0.25%) after surgery using ultrasonographic guidance.

ELIGIBILITY:
Inclusion Criteria:

* 75 patients, aged between 21- 80 years old, of both sex American society of Anesthesiology I - III scheduled for total hip replacement surgery.

Exclusion Criteria:

* Patient refusal.
* Coagulopathy
* Spinal deformities
* Peripheral neuropathy; sensory disorders in the leg requiring surgery and chronic pain.
* Mental dysfunction, psychiatric illnesses and cognitive dysfunction.
* History of drug abuse &chronic analgesic use

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine consumption | Baseline
  Total Morphine consumption in the first 24 h of the post-operative period .

SECONDARY OUTCOMES:
Postoperative pain score | Baseline
  • Postoperative pain will be assessed by VAS (score for the severity of pain in the range 0-10, where 0 = no pain and 10 = severe pain) at 2,4,6,12,18,24 hours. If the VAS is 4 or more, 3 mg of intravenous morphine will be given as a rescue analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: YASSER M RAGHEB, PROF, Study Chair — TANYAU
Locations (1):
- Tanata university hospital, Tanta, Egypt

REFERENCES:
- [Background] Singh JA, Lewallen D. Predictors of pain and use of pain medications following primary Total Hip Arthroplasty (THA): 5,707 THAs at 2-years and 3,289 THAs at 5-years. BMC Musculoskelet Disord. 2010 May 13;11:90. doi: 10.1186/1471-2474-11-90. PMID 20462458
- [Background] Abduallah MA, Ahmed SA, Abdelghany MS. The effect of post-operative ultrasound-guided transmuscular quadratus lumborum block on post-operative analgesia after hip arthroplasty in elderly patients: A randomised controlled double-blind study. Indian J Anaesth. 2020 Oct;64(10):887-893. doi: 10.4103/ija.IJA_275_20. Epub 2020 Oct 1. PMID 33437078

DOCUMENTS (1):
  • Study Protocol (2021-07-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT05465967/Prot_001.pdf